CLINICAL TRIAL: NCT00496769
Title: Apixaban Versus Acetylsalicylic Acid (ASA) to Prevent Stroke in Atrial Fibrillation Patients Who Have Failed or Are Unsuitable for Vitamin K Antagonist Treatment: A Randomized Double-blind Trial
Brief Title: A Phase III Study of Apixaban in Patients With Atrial Fibrillation
Acronym: AVERROES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV185-048
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Experimental)
  Interventions: Drug: Apixaban
- Acetylasalicylic acid (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Apixaban — Tablets, oral, 5 mg (2.5 mg in patients meeting any 2 of the following criteria: 80 years of age and older, weight of 60 kilograms or less, and a serum creatinine level of 1.5 mg/dL or higher), twice daily, up to 156 weeks
  Other Names: BMS-562247
  Arms: Apixaban
Drug: Acetylsalicylic acid — Tablets, oral, 81-324 mg, once daily, up to 156 weeks
  Arms: Acetylasalicylic acid

SUMMARY:
The purpose of this clinical research study is to determine whether apixaban is more effective than acetylsalicylic acid in the prevention of strokes associated with patients with atrial fibrillation. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
An optional Long-term Open-label Extension Phase of treatment with apixaban will be provided for qualifying participants following the conclusion of the double-blind phase

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female
* Age of 50 years or older
* Permanent, paroxysmal, or persistent atrial fibrillation (at screening or within 6 months prior to enrollment) documented by 12-lead electrocardiogram)
* At least 1 of the following risk factors for stroke:

  * Prior stroke or transient ischemic attack
  * Age of 75 years or older
  * Arterial hypertension on treatment
  * Diabetes mellitus
  * Heart failure (New York Health Authority Class 2 or greater at time of enrollment)
  * Left ventricular ejection fraction of 35% or less, documented within 6 months of enrollment
  * Peripheral arterial disease (previous arterial revascularization, limb or foot amputation, or current intermittent claudication with ankle-arm systolic blood pressure ratio <0.9)
* Not currently receiving vitamin K antagonist therapy for 1 of the following reasons:

  * Previous vitamin K antagonist therapy demonstrated as unsuitable and discontinued
  * Vitamin K antagonist therapy not previously used but expected unsuitable

Key Exclusion Criteria:

* Women who are pregnant or breast feeding
* Women of child bearing potential who are unwilling to meet the study requirements for pregnancy testing or are unwilling or unable to use an acceptable method to avoid pregnancy
* Atrial fibrillation due to reversible causes, such as thyrotoxicosis or pericarditis
* Valvular disease requiring surgery
* Planned ablation procedure for atrial fibrillation to be performed within 3 months
* Conditions other than atrial fibrillation that require chronic anticoagulation (such as, prosthetic mechanical heart valve, venous thromboembolism)
* Patients with serious bleeding in the last 6 months or at high risk for bleeding, including but not limited to those with:

  * Active peptic ulcer disease
  * Platelet count <100,000/mm^3 or hemoglobin <10g/dL
  * Recent stroke (within 10 days)
  * Documented hemorrhagic tendencies or blood dyscrasias
* Current alcohol or drug abuse or psychosocial reasons that make study participation impractical
* Severe comorbid condition with life expectancy <1 year
* Severe renal insufficiency; any patient with a serum creatinine level >2.5 mg/dL or a calculated creatinine clearance <25 mL/min is excluded
* Alanine transaminase or aspartate aminotransferase levels >2 times upper limit of normal (ULN) or a total bilirubin level >1.5 times ULN (unless an alternative causative factor [such as Gilbert's syndrome] is identified)
* Allergy or adverse reaction to acetylsalicylic acid
* Required treatment with a thienopyridine (clopidogrel or ticlopidine)
* Prisoners or participants who are compulsory detained (involuntarily incarcerated)
* Use of an investigational drug or device within the past 30 days or prior randomization into an apixaban clinical study
* Patients who are compulsorily detained for treatment for a psychiatric or physical illness

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6421 (Actual)
Dates: Start 2007-08-31 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (395):
- United States (69):
  - Mobile Heart Specialists, Pc, Mobile, Alabama
  - Southwest Heart, Tucson, Arizona
  - Cardiology Consultants Of Orange County Med. Group Inc, Anaheim, California
  - Kaiser Permanente Medical Center, West Los Angeles, Los Angeles, California
  - Desert Med Grp Inc, Dba Desert Oasis Healthcare Med Group, Palm Springs, California
  - Yogesh K. Paliwal Md, Pomona, California
  - San Diego Managed Care Group, Poway, California
  - University Of California, San Diego, San Diego, California
  - Santa Rosa Cardiology, Santa Rosa, California
  - North County Internal Medicine, Vista, California
  - Cardiology Associates Of New Haven,Pc, Guilford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Bay Pines Va Healthcare System, Bay Pines, Florida
  - Research Alliance, Inc., Clearwater, Florida
  - The Heart & Vascular Institute Of Florida, Clearwater, Florida
  - Kim A. Klancke, Md, Daytona Beach, Florida
  - The Heart Group Pl, Fort Myers, Florida
  - St. Vincent'S Ambulatory Care, Inc, Jacksonville, Florida
  - Baptist Heart Specialists, Jacksonville Beach, Florida
  - Michael F. Lesser, Md, Facc Osler Medical Inc., Melbourne, Florida
  - Cardiovascular Center Of Sarasota, Sarasota, Florida
  - The Broward Heart Group, Pa, Tamarac, Florida
  - Southeast Regional Research Group, Columbus, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - Fox Valley Clinical Research Center, Llc, Aurora, Illinois
  - North Chicago Va Medical Center, North Chicago, Illinois
  - Indiana Heart Physicians, Inc., Indianapolis, Indiana
  - The Care Group, Llc, Indianapolis, Indiana
  - Hutchinson Clinic, Pa, Hutchinson, Kansas
  - Dr. Jeffrey Chen, Lafayette, Louisiana
  - Peninsula Cardiology Associates, P.A., Salisbury, Maryland
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Great Lakes Heart Center Of Alpena, Alpena, Michigan
  - Henry Ford Hospital K-15, Detroit, Michigan
  - Michigan Heart And Vascular Specialists, Petoskey, Michigan
  - Academic Cardiology Associates, Rochester Hills, Michigan
  - Tupelo Neurology Clinic, Pa, Tupelo, Mississippi
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - University Of Missouri, Columbia, Missouri
  - Glacier View Cardiology, Pc, Kalispell, Montana
  - Hunterdon Cardiovascular Associates, Flemington, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - Nyu Hudson Valley Cardiology, Cortlandt Manor, New York
  - Long Island Heart Associates, Mineola, New York
  - Dr William Kufs, Saratoga Springs, New York
  - Capital Cardiology Associates, Troy, New York
  - Terry V. Arnold, Md, Lexington, North Carolina
  - Pinehurst Medical Clinic, Inc, Pinehurst, North Carolina
  - Sanford Cardiology, Sanford, North Carolina
  - Ira R. Friedlander, M.D., Canton, Ohio
  - Davis Heart & Lung Research Institute, Columbus, Ohio
  - Integris Cardiovascular Physicians, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Oregon Medical Group - Clinical Research, Eugene, Oregon
  - Hillsboro Cardiology Pc, Hillsboro, Oregon
  - The Portland Clinic, Llp, Portland, Oregon
  - Comprehensive Cardiology Consultants, Langhorne, Pennsylvania
  - Grand View - Lehigh Valley Health Services, Sellersville, Pennsylvania
  - West Chester Cardiology, West Chester, Pennsylvania
  - Cardiology Consultants Of Philadelphia, Yardley, Pennsylvania
  - Lowcountry Medical Group, Llc, Beaufort, South Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - Internal Medicine Of Greer, Greer, South Carolina
  - Knoxville Heart Group, Knoxville, Tennessee
  - Sentara York Clinical Research, Norfolk, Virginia
  - Roanoke Heart Institute, Plc, Roanoke, Virginia
  - Salem Veterans Administration Medical Center, Salem, Virginia
  - Walla Walla Clinic, Walla Walla, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Argentina (19):
  - Local Institution, Adrogué, Buenos Aires
  - Local Institution, Autonoma Buenos Aires, Buenos Aires
  - Local Institution, Bahía Blanca, Buenos Aires
  - Local Institution, Coronel Suárez, Buenos Aires
  - Local Institution, Haedo, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Merlo, Buenos Aires
  - Local Institution, Ramos Mejía, Buenos Aires
  - Local Institution, San Francisco, Córdoba Province
  - Local Institution, San Salvador de Jujuy, Jujuy Province
  - Local Institution, Zárate, Provincia Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
  - Local Institution, Buenos Aires
  - Local Institution, Corrientes
  - Local Institution, Córdoba
  - Local Institution, Salta
  - Local Institution, Santa Fe
- Australia (10):
  - Local Institution, Coffs Harbour, New South Wales
  - Local Institution, Concord, New South Wales
  - Local Institution, Gosford, New South Wales
  - Local Institution, Kingswood, New South Wales
  - Local Institution, Auchenflower, Queensland
  - Local Institution, Kippa-Ring, Queensland
  - Local Institution, Milton, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Geelong, Victoria
  - Local Institution, Joondalup, Western Australia
- Austria (4):
  - Local Institution, Graz
  - Local Institution, Linz
  - Local Institution, Oberpullendorf
  - Local Institution, Salzburg
- Belgium (8):
  - Local Institution, Aalst
  - Local Institution, Brasschaat
  - Local Institution, Brussels
  - Local Institution, De Pinte
  - Local Institution, Genk
  - Local Institution, Huy
  - Local Institution, Roeselare
  - Local Institution, Turnhout
- Brazil (18):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Uberaba, Minas Gerais
  - Local Institution, Campina Grande do Sul, Paraná
  - Local Institution, Curitiba, Paraná
  - Local Institution, Maringá, Paraná
  - Local Institution, Belém, Pará
  - Local Institution, Natal, Rio Grande do Norte
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Blumenau, Santa Catarina
  - Local Institution, São José, Santa Catarina
  - Local Institution, Botucatu, São Paulo
  - Local Institution, Campinas, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, San Jose- Do Rio Preto, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (22):
  - Local Institution, New Westminster, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Brampton, Ontario
  - Local Institution, Burlington, Ontario
  - Local Institution, Cambridge, Ontario
  - Local Institution, Greater Sudbury, Ontario
  - Local Institution, Grimsby, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Weston, Ontario
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Saint Georges Beauce, Quebec
  - Local Institution, Saint-Jérôme, Quebec
  - Local Institution, Saint-Lambert, Quebec
  - Local Institution, Terrebonne, Quebec
  - Local Institution, Westmount, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Chile (6):
  - Local Institution, Osorno, Los Lagos Region
  - Local Institution, Valdivia, Los Ríos Region
  - Local Institution, Temuco, Región de la Araucanía
  - Local Institution, Victoria, Región de la Araucanía
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Santiago, Santiago Metropolitan
- China (10):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Shijiazhuang, Hebei
  - Local Institution, Wuhan, Hubei
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Dalian, Liaoning
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Qingdao, Shandong
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
- Colombia (5):
  - Local Institution, Medellín, Antioquia
  - Local Institution, Barranquilla, Atlántico
  - Local Institution, Bucaramanga, Santander Department
  - Local Institution, Cali, Valle del Cauca Department
  - Local Institution, Bogotá
- Czechia (13):
  - Local Institution, Brno
  - Local Institution, Havirov - Mesto
  - Local Institution, Jindřichův Hradec
  - Local Institution, Kladno
  - Local Institution, Kroměříž
  - Local Institution, Městec Králové
  - Local Institution, Ostrava
  - Local Institution, Písek
  - Local Institution, Prague
  - Local Institution, Přelouč
  - Local Institution, Příbram
  - Local Institution, Slaný
  - Local Institution, Ústí nad Orlicí
- Denmark (3):
  - Local Institution, Arhus C
  - Local Institution, Esbjerg
  - Local Institution, Frederiksberg
- Finland (5):
  - Local Institution, Espoo
  - Local Institution, Helsinki
  - Local Institution, Jyväskylä
  - Local Institution, Kuopio
  - Local Institution, Tampere
- France (8):
  - Local Institution, Abbeville
  - Local Institution, Albi
  - Local Institution, Cholet
  - Local Institution, Grenoble
  - Local Institution, Langres
  - Local Institution, Paris
  - Local Institution, Sisteron
  - Local Institution, Toulon
- Germany (18):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Cologne
  - Local Institution, Essen
  - Local Institution, Frankfurt am Main
  - Local Institution, Halle
  - Local Institution, Hamburg
  - Local Institution, Heidelberg
  - Local Institution, Kassel
  - Local Institution, Leipzig
  - Local Institution, Magdeburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, Papenburg
  - Local Institution, Regensburg
  - Local Institution, Riesa
  - Local Institution, Witten
  - Local Institution, Wolmirstedt
- Greece (3):
  - Local Institution, Athens
  - Local Institution, Larissa
  - Local Institution, Thebes
- Hong Kong (3):
  - Local Institution, Shatin, NEW Territories
  - Local Institution, Chai Wan
  - Local Institution, Hong Kong
- India (18):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Banglore, Karnataka
  - Local Institution, Mysore, Karnataka
  - Local Institution, Mumbai, Maharashtra
  - Local Institution, Nagpur, Maharashtra
  - Local Institution, Nashik, Maharashtra
  - Local Institution, Pune, Maharashtra
  - Local Institution, Dhantoli, Nagpur
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Lucknow, Uttar Pradesh
  - Local Institution, Ahmedabad
  - Local Institution, Bangalore
  - Local Institution, Bikaner
  - Local Institution, Indore
  - Local Institution, Jaipur
  - Local Institution, Kottayam
  - Local Institution, Pune
- Indonesia (9):
  - Local Institution, Malang, East Java
  - Local Institution, Bandung
  - Local Institution, Denpasar
  - Local Institution, Jakarta
  - Local Institution, Jakarta Timur
  - Local Institution, Padang
  - Local Institution, Palembang
  - Local Institution, Surabaya
  - Local Institution, Yogyakarta
- Israel (10):
  - Local Institution, Afula
  - Local Institution, Ashkelon
  - Local Institution, Giv‘atayim
  - Local Institution, Hadera
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Nazareth
  - Local Institution, Petah Tikva
  - Local Institution, Safed
  - Local Institution, Tel Aviv
- Italy (9):
  - Local Institution, Ascoli Piceno
  - Local Institution, Chieti
  - Local Institution, Genova
  - Local Institution, Isernia
  - Local Institution, Lido di Camaiore
  - Local Institution, Palermo
  - Local Institution, Perugia
  - Local Institution, San Daniele de Friuli (ud)
  - Local Institution, Sassari
- Malaysia (5):
  - Local Institution, Johor Bahru, Johor
  - Local Institution, Cheras, Kuala Lumpur
  - Local Institution, Pulau Pinang, Pulau Pinang
  - Local Institution, Kuching, Sarawak
  - Local Institution, Kuala Lumpur
- Mexico (15):
  - Local Institution, Acapulco de Juárez, Guerrero
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, San Luis Potosi, Slp, San Luis Potosí
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Hermosillo, Sonora
  - Local Institution, Ciudad López Mateos, State of Mexico
  - Local Institution, Jalapa, Veracruz
  - Local Institution, Aguascalientes
  - Local Institution, Chihuahua City
  - Local Institution, Durango
  - Local Institution, Querétaro
  - Local Institution, San Luis Potosí City
- Norway (3):
  - Local Institution, Fyllingsdal
  - Local Institution, Kongsberg
  - Local Institution, Oslo
- Philippines (8):
  - Local Institution, Naga, Camarines SUR
  - Local Institution, Biñan, Laguna
  - Local Institution, Iligan City, Lanao DEL Norte
  - Local Institution, Cagayan de Oro
  - Local Institution, Cavite
  - Local Institution, City of Muntinlupa
  - Local Institution, Laoag
  - Local Institution, Manila
- Poland (21):
  - Local Institution, Częstochowa
  - Local Institution, Elblag
  - Local Institution, Gdynia
  - Local Institution, Gliwice
  - Local Institution, Gniewkowo
  - Local Institution, Grodzisk Mazowiecki
  - Local Institution, Inowrocław
  - Local Institution, Kielce
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Piotrkow Trybunalski
  - Local Institution, Poznan
  - Local Institution, Puławy
  - Local Institution, Płock
  - Local Institution, Siemianowice Śląskie
  - Local Institution, Skierniewice
  - Local Institution, Tarnów
  - Local Institution, Warsaw
  - Local Institution, Węgrów
  - Local Institution, Zabrze
  - Local Institution, Żarów
- Russia (19):
  - Local Institution, Kaluga, Anenki
  - Local Institution, Barnaul
  - Local Institution, Chelyabinsk
  - Local Institution, Kazan'
  - Local Institution, Kemerovo
  - Local Institution, Krasnodar
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Novosibirsk
  - Local Institution, Perm
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Saratov
  - Local Institution, Tomsk
  - Local Institution, Tver'
  - Local Institution, Tyumen
  - Local Institution, Yaroslavl
  - Local Institution, Yekaterinburg
- Local Institution, Singapore, Singapore
- South Africa (7):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Alberton, Gauteng
  - Local Institution, Bellville, Cape Town, Western Cape
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Somerset West, Western Cape
  - Local Institution, Worcester, Western Cape
  - Local Institution, Pretoria
- South Korea (8):
  - Local Institution, Goyang-si, Gyeonggi-do
  - Local Institution, Guri-si, Gyeonggi-do
  - Local Institution, Seongnam-si, Gyeonggi-do
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Gwangju
  - Local Institution, Seoul
- Spain (6):
  - Local Institution, Torrevieja, Alicante
  - Local Institution, L'Hospitalet de Llobregat, Barcelona
  - Local Institution, Lugo, Galicia
  - Local Institution, Albacete
  - Local Institution, Madrid
  - Local Institution, Valencia
- Sweden (4):
  - Local Institution, Gothenburg
  - Local Institution, Mölndal
  - Local Institution, Stockholm
  - Local Institution, Uppsala
- Taiwan (4):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
- Turkey (Türkiye) (3):
  - Local Institution, Isparta
  - Local Institution, Istanbul
  - Local Institution, Kırıkkale
- Ukraine (4):
  - Local Institution, Dnipropetrovsk
  - Local Institution, Donetsk
  - Local Institution, Kharkiv
  - Local Institution, Kyiv
- United Kingdom (17):
  - Local Institution, Aberdeen, Aberdeenshire
  - Local Institution, Chesterfield, Derbyshire
  - Local Institution, Basildon, Essex
  - Local Institution, Romford, Essex
  - Local Institution, Kirkcaldy, Fife
  - Local Institution, London, Greater London
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Blackpool, Lancashire
  - Local Institution, Northampton, Northamptonshire
  - Local Institution, Worksop, Nottinghamshire
  - Local Institution, Craigavon, Portadown
  - Local Institution, Paisley, Renfrewshire
  - Local Institution, Barnsley, South Yorkshire
  - Local Institution, Larbert, Stirlingshire
  - Local Institution, Newcastle Upon, Tyne and Wear
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Chichester, West Sussex

REFERENCES:
- [Derived] Jamieson MJ, Byon W, Dettloff RW, Crawford M, Gargalovic PS, Merali SJ, Onorato J, Quintero AJ, Russ C. Apixaban Use in Obese Patients: A Review of the Pharmacokinetic, Interventional, and Observational Study Data. Am J Cardiovasc Drugs. 2022 Nov;22(6):615-631. doi: 10.1007/s40256-022-00524-x. Epub 2022 May 16. PMID 35570249
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Bhagirath VC, Eikelboom JW, Hirsh J, Coppens M, Ginsberg J, Vanassche T, Yuan F, Chan N, Yusuf S, Connolly SJ. Apixaban-Calibrated Anti-FXa Activity in Relation to Outcome Events and Clinical Characteristics in Patients with Atrial Fibrillation: Results from the AVERROES Trial. TH Open. 2017 Dec 12;1(2):e139-e145. doi: 10.1055/s-0037-1613679. eCollection 2017 Jul. PMID 31249919
- [Derived] Ng KH, Shestakovska O, Connolly SJ, Eikelboom JW, Avezum A, Diaz R, Lanas F, Yusuf S, Hart RG. Efficacy and safety of apixaban compared with aspirin in the elderly: a subgroup analysis from the AVERROES trial. Age Ageing. 2016 Jan;45(1):77-83. doi: 10.1093/ageing/afv156. Epub 2015 Nov 19. PMID 26590293
- [Derived] Hohnloser SH, Shestakovska O, Eikelboom J, Franzosi MG, Tan RS, Zhu J, Yusuf S, Connolly SJ. The effects of apixaban on hospitalizations in patients with different types of atrial fibrillation: insights from the AVERROES trial. Eur Heart J. 2013 Sep;34(35):2752-9. doi: 10.1093/eurheartj/eht292. Epub 2013 Jul 25. PMID 23892201
- [Derived] Lip GY, Connolly S, Yusuf S, Shestakovska O, Flaker G, Hart R, Lanas F, Xavier D, Eikelboom J; ERROES Investigators. Modification of outcomes with aspirin or apixaban in relation to CHADS(2) and CHA(2)DS(2)-VASc scores in patients with atrial fibrillation: a secondary analysis of the AVERROES study. Circ Arrhythm Electrophysiol. 2013 Feb;6(1):31-8. doi: 10.1161/CIRCEP.112.975847. Epub 2013 Feb 6. PMID 23390125
- [Derived] Flaker GC, Eikelboom JW, Shestakovska O, Connolly SJ, Kaatz S, Budaj A, Husted S, Yusuf S, Lip GY, Hart RG. Bleeding during treatment with aspirin versus apixaban in patients with atrial fibrillation unsuitable for warfarin: the apixaban versus acetylsalicylic acid to prevent stroke in atrial fibrillation patients who have failed or are unsuitable for vitamin K antagonist treatment (AVERROES) trial. Stroke. 2012 Dec;43(12):3291-7. doi: 10.1161/STROKEAHA.112.664144. Epub 2012 Oct 2. PMID 23033347
- [Derived] Diener HC, Eikelboom J, Connolly SJ, Joyner CD, Hart RG, Lip GY, O'Donnell M, Hohnloser SH, Hankey GJ, Shestakovska O, Yusuf S; AVERROES Steering Committee and Investigators. Apixaban versus aspirin in patients with atrial fibrillation and previous stroke or transient ischaemic attack: a predefined subgroup analysis from AVERROES, a randomised trial. Lancet Neurol. 2012 Mar;11(3):225-31. doi: 10.1016/S1474-4422(12)70017-0. Epub 2012 Feb 1. PMID 22305462
- [Derived] Connolly SJ, Eikelboom J, Joyner C, Diener HC, Hart R, Golitsyn S, Flaker G, Avezum A, Hohnloser SH, Diaz R, Talajic M, Zhu J, Pais P, Budaj A, Parkhomenko A, Jansky P, Commerford P, Tan RS, Sim KH, Lewis BS, Van Mieghem W, Lip GY, Kim JH, Lanas-Zanetti F, Gonzalez-Hermosillo A, Dans AL, Munawar M, O'Donnell M, Lawrence J, Lewis G, Afzal R, Yusuf S; AVERROES Steering Committee and Investigators. Apixaban in patients with atrial fibrillation. N Engl J Med. 2011 Mar 3;364(9):806-17. doi: 10.1056/NEJMoa1007432. Epub 2011 Feb 10. PMID 21309657
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 6421 patients were enrolled in the study. Of these, 5598 were randomized (2807 to apixaban and 2791 to acetylsalicylic acid). Most (435) of the patients who were not randomized (823) no longer met study criteria. Of those randomized, 5578 received treatment (2798 with apixaban, and 2780 with acetylsalicylic acid).
Groups:
- Apixaban, 2.5 or 5 mg Twice Daily: Patients received 5 mg of apixaban twice daily. Participants who fulfilled any 2 of the following criteria at baseline received apixaban, 2.5 mg twice daily: age older than 80 years, body weight of 60 kg or less, Serum creatinine level ≥1.5 mg/dL. Participants randomized to the 2.5 mg twice daily dose of apixaban continued on this dose throughout the study even if they no longer fulfilled the previous criteria.
- Acetylsalicylic Acid, 81-324 mg Once Daily: Patients received 81 to 324 mg of acetylsalicylic acid once daily, with dosage based on investigator discretion Participants who completed the double-blind treatment period and met eligibility criteria had the option of enrolling in the Long Term Open Label Extension to receive open-label apixaban.
- Open Label Apixaban: Participants who completed the double-blind treatment period and met eligibility criteria had the option of enrolling in the Long Term Open Label Extension to receive open-label apixaban.
Period: Double Blind
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily | Open Label Apixaban
Started | 2807 (Randomized) | 2791 (Randomized) | 0
Received Treatment | 2798 | 2708 | 0
Completed | 2249 | 2142 | 0
Not Completed | 558 | 649 | 0
Not completed — >=1 reason assigned per patient | 558 | 649 | 0
Period: Open Label
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily | Open Label Apixaban
Started | 0 | 0 | 3275
Completed | 0 | 0 | 2264
Not Completed | 0 | 0 | 1011
Not completed — >=1 reason assigned per patient | 0 | 0 | 1011

BASELINE CHARACTERISTICS:
Groups:
- Acetylsalicylic Acid, 81-324 mg Once Daily: Patients received 81 to 324 mg of acetylsalicylic acid once daily, with dosage based on investigator discretion
- Total: Total of all reporting groups
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily | Total
Number analyzed (Participants) | 2807 | 2791 | 5598
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (9.44) | 70.0 (9.71) | 69.9 (9.58)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 855 | 865 | 1720
  >=65 but <75 years | 1049 | 938 | 1987
  >=75 years | 903 | 988 | 1891
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1147 | 1174 | 2321
  Male | 1660 | 1617 | 3277
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 12
  Asian | 541 | 544 | 1085
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 10 | 26 | 36
  White | 2221 | 2178 | 4399
  Other | 26 | 36 | 62
Number of Participants by Number of Risk Factors for Stroke [Count of Participants; unit: Participants]
  1 or fewer | 1085 | 1077 | 2162
  2 or more | 1722 | 1714 | 3436
Number of Participants With Risk Factors for Stroke [Count of Participants; unit: Participants] — NYHA=New York Health Authority; LVEF=left ventricular ejection fraction
  Participants
    Age of 75 years or older | 903 | 988 | 1891
    Prior stroke or transient ischemic attack | 390 | 374 | 764
    Heart failure (NYHA class ≥2) or LVEF ≤35% | 961 | 926 | 1887
    Diabetes mellitus | 536 | 559 | 1095
    Hypertension requiring pharmacologic treatment | 2408 | 2429 | 4837
    Peripheral artery disease | 66 | 78 | 144

OUTCOME MEASURES:

1. Primary Outcome: Event Rate of Stroke/Systemic Embolism During the Intended-treatment Period
Description: Event rate=percent of participants with an event divided by the total participants in the arm. Intended-treatment period=date of randomization to the efficacy cutoff date, which was to be the date on which at least 226 unrefuted original primary efficacy events occurred (date revised to May 28, 2010 following cessation of study for superior efficacy.)
Time Frame: Randomization to efficacy cutoff date of May 28, 2010 (date revised following cessation of study for superior efficacy)
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of events
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2807 | 2791
Percentage of events | 1.62 | 3.63
Statistical Analysis 1: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Superiority; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.32 to 0.62]

2. Secondary Outcome: Event Rate for the Composite of Stroke of Any Type, Systemic Embolism, Myocardial Infarction, or Vascular Death During the Double-blind Treatment Period
Description: Event rate=percent of participants with an event divided by the total participants in the arm.
Time Frame: Randomization to efficacy cutoff date of May 28, 2010 (date revised following cessation of study for superior efficacy)
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of events per year
Groups:
- Apixaban, 2.5 or 5 mg Twice Daily: Patients received 5 mg of apixaban twice daily. Participants who fulfilled any 2 of the following criteria at baseline received apixaban, 2.5 mg twice daily: age older than 80 years, body weight of 60 kg or less, Serum creatinine level ≥1.5 mg/dL. Participants randomized to the 2.5 mg twice daily dose of apixaban continued on this dose throughout the study even if they no longer fulfilled the previous criteria.
  Participants who completed the double-blind treatment period and met eligibility criteria had the option of enrolling in the Long Term Open Label Extension to receive open-label apixaban.
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2807 | 2791
Percentage of events per year | 4.21 | 6.35
Statistical Analysis 1: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Superiority; p = 0.00026, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.53 to 0.83] — Vascular death

3. Secondary Outcome: Event Rate of All-cause Death; Net Clinical Benefit-Composite of Stroke, Systemic Embolism, Myocardial Infarction, Vascular Death, and Major Bleeding; and Vascular Death
Description: Event rate=percent of participants with an event divided by the total participants in the arm.
Time Frame: Randomization to efficacy cutoff date of May 28, 2010 (date revised following cessation of study for superior efficacy)
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of events per year
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2807 | 2791
Percentage of events per year
  All-cause death (n=111, 140) | 3.51 | 4.42
  Net clinical benefit (n=163, 220) | 5.23 | 7.13
  Vascular death (n=84, 96) | 2.65 | 3.03
Statistical Analysis 1: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Superiority; p = 0.06782, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.62 to 1.02] — All-cause death
Statistical Analysis 2: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Superiority; p = 0.00280, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.60 to 0.90] — Composite endpoint of major vascular events and major bleeding-net clinical benefit
Statistical Analysis 3: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Superiority; p = 0.36586, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.65 to 1.17] — Vascular death

4. Secondary Outcome: Event Rates for Major Bleeding, Major or Clinically Relevant Nonmajor (CNRM) Bleeding, and All Bleeding in the Double-blind Period
Description: Event rate=percent of participants with an event divided by the total participants in the arm.
Time Frame: First dose of study drug (Day 1) to the earlier of a patient's discontinuation of double-blind study drug or the attainment of at least 226 primary efficacy events up to May 28, 2010
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of events per year
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2798 | 2780
Percentage of events per year
  Major bleeding | 1.41 | 0.92
  Major or CRNM bleeding | 4.46 | 3.24
  All bleeding | 10.85 | 8.32
Statistical Analysis 1: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Other; p = 0.0716, Log Rank; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.96 to 2.45] — Major bleeding
Statistical Analysis 2: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Other; p = 0.0017, Log Rank; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [1.10 to 1.53] — All bleeding
Statistical Analysis 3: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Other; p = 0.0144, Log Rank; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [1.07 to 1.78] — Major or CNRM bleeding

5. Secondary Outcome: Rate of Unrefuted Bleeding From First Dose of Double-blind Study Drug to First Occurence of Unrefuted Bleeding During the Double-blind Treatment Period
Description: Event rate=percent of participants with an event divided by the total participants in the arm.
Time Frame: Day 1 to first bleeding event up to efficacy cutoff date of May 28, 2010 (date revised following cessation of study for superior efficacy)
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of events per year
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2798 | 2780
Percentage of events per year | 10.85 | 8.32
Statistical Analysis 1: Comparison: Apixaban, 2.5 or 5 mg Twice Daily vs Acetylsalicylic Acid, 81-324 mg Once Daily; Test type: Other; p = 0.0017, Log Rank; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [1.10 to 1.53]

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events (AEs), Bleeding AEs, Discontinuations Due to AEs, and Death as Outcome
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: First dose of study drug (Day 1) to 30 days after last dose of blinded study drug
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2798 | 2780
Participants
  AEs | 1833 | 1925
  SAEs | 657 | 804
  Bleeding AEs | 281 | 259
  Discontinuations due to AE | 266 | 362
  Deaths | 91 | 115

7. Secondary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Marked Abnormality
Description: BL=baseline, LLN=lower limit of normal, ULN=upper limit of normal. Hemoglobin (g/dL), low: BL>2 or value ≤8; hematocrit(%), low: <0.75*BL; erythrocytes (*10^6 cells/μL), low: <0.75*BL; platelet count (*10^9 cells/L),low: <100*10^9 cells/L; leukocytes (*10^3 cells/μL), low if <0.8*BL and BL<LLN or <LLN and BL >ULN or <0.75*LLN when BL is missing or LLN ≤BL≤ ULN, high if >1.2*BL and BL>ULN or >ULN when BL and BL<LLN or >1.25*ULN when BL is missing or LLN≤BL≤ULN; neutrophils (absolute), low: <1.0*10^3 cells/μL; eosinophils (absolute), high: >0.750*10^3 cells/μL; basophils (absolute), high: >0.4*10^3 cells/μL; monocytes (absolute), high: 2*10^3 cells/μL; lymphocytes (absolute), low if <0.75*10^3 cells/μL, high if >7.50*10^3 cells/μL; ALP (U/L), high: 2*ULN; AST (U/L), high: 3*ULN; AST (U/L), high: 3*ULN; bilirubin, total (mg/dL), high: >2*ULN; bilirubin, direct (mg/dL), high: 1.5*ULN; BUN (mg/dL), high:>2*ULN; creatinine (mg/dL), high: >1.5*ULN.
Time Frame: First dose of study drug (Day 1) to 30 days after last dose of blinded study drug
Population: Participants who received at least 1 dose of study drug. n=number evaluable
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2798 | 2780
Participants
  Hemoglobin, low (n=1956, 1893) | 131 | 120
  Hemoglobin, high (n=1956, 1893) | 0 | 0
  Hematocrit, low (n=1728, 1687) | 13 | 9
  Hematocrit, high (n=1728, 1687) | 0 | 0
  Erythrocytes, low (n=1728, 1687) | 12 | 12
  Erythrocytes, high (n=1728, 1687) | 0 | 0
  Platelet count, low (n=2148, 2098) | 7 | 10
  Platelet count, high (n=2148, 2098) | 0 | 0
  Leukocytes, low (n=1738, 1698) | 12 | 14
  Leukocytes, high (n=1738, 1698) | 14 | 18
  Neutrophils (absolute), low (n=2170, 2138) | 2 | 1
  Neutrophils (absolute), high (n=2170, 2138) | 0 | 0
  Eosinophils (absolute), low (n=2170, 2138) | 0 | 0
  Eosinophils (absolute), high (n=2170, 2138) | 48 | 68
  Basophils (absolute), low (n=2170, 2138) | 0 | 0
  Basophils (absolute), high (n=2170, 2138) | 0 | 0
  Monocytes (absolute), low (n=2170, 2138) | 0 | 0
  Monocytes (absolute), high (n=2170, 2138) | 0 | 2
  Lymphocytes (absolute), low (n=2170, 2138) | 52 | 62
  Lymphocytes (absolute), high (n=2170, 2138) | 4 | 5
  Alkaline phosphatase (ALP), low (n=2781, 2758) | 0 | 0
  ALP, high (n=2781, 2758) | 34 | 27
  Aspartate phosphatase (AST), low (n=2779, 2753) | 0 | 0
  AST, high (n=2779, 2753) | 28 | 33
  Alanine aminotransferase (ALT), low (n=2779, 2753) | 0 | 0
  ALT, high (n=2779, 2753) | 23 | 31
  Bilirubin (total), low (n=2781, 2758) | 0 | 0
  Bilirubin (total), high (n=2781, 2758) | 30 | 43
  Bilirubin (direct), low (n=2773, 2750) | 0 | 0
  Bilirubin (direct), high (n=2773, 2750) | 241 | 248
  Blood urea nitrogen (BUN), low (n=2201, 2172) | 0 | 0
  BUN, high (n=2201, 2172) | 42 | 50
  Creatinine, low (n=2209, 2178) | 0 | 0
  Creatinine, high (n=2209, 2178) | 67 | 71

8. Secondary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Marked Abnormality (Continued)
Description: LLN=lower limit of normal; ULN=upper limit of normal; BL=baseline. Sodium, serum (mEq/L):low if <0.95*BL and BL<LLN or <LLN and BL>ULN or <0.95*LLN when BL missing or LLN ≤BL≤ULN, high if >1.05*BL and BL>ULN or >ULN and BL<LLN or >1.05*ULN when BL missing or LLN≤BL≤ULN; potassium(mEq/L):low if <0.90*BL and BL<LLN or <LLN and BL>ULN or <0.90*LLN if BL missing or LLN≤BL≤ULN, high if >1.10*BL and BL>ULN or>ULN and BL<LLN or >1.10*ULN when BL missing or LLN≤BL≤ULN; chloride(mEq/L):low if <0.90*BL and BL<LLN or <LLN and BL>ULN or <0.90*LLN if BL missing or LLN≤BL ≤ULN, high if >1.10*BL and BL>ULN or >ULN and BL<LLN or >1.10* ULN if BL missing or LLN≤BL≤ULN; calcium(mg/dL):low if <0.75*BL and BL<LLN or <LLN and BL>ULN or <0.80*LLN if BL missing or LLN≤BL≤ULN, high if >1.25*BL and BL>ULN or >ULN if BL<LLN or >1.20*ULN if BL missing or LLN≤BL≤ULN ; bicarbonate(mEq/L):low if <0.75*BL when BL<LLN or <LLN when BL>ULN or <0.75*LLN if BL missing or LLN≤BL≤ULN, high if >1.25*BL when BL>ULN or >ULN
Time Frame: First dose of study drug (Day 1) to 30 days after last dose of blinded study drug
Population: Participants who received at least 1 dose of study drug. n=number evaluable
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2798 | 2780
Participants
  Sodium (serum), low (n=1768, 1740) | 2 | 6
  Sodium (serum), high (n=1768, 1740) | 1 | 2
  Potassium (serum), low (n=1763, 1737) | 6 | 8
  Potassium (serum), high (n=1763, 1737) | 20 | 28
  Chloride (serum), low (n=1768, 1740) | 0 | 3
  Chloride (serum), high (n=1768, 1740) | 0 | 1
  Calcium (total), low (n=106, 109) | 0 | 0
  Calcium (total), high (n=106, 109) | 0 | 0
  Bicarbonate, low (n=1664, 1619) | 0 | 0
  Bicarbonate, high (n=1664, 1619) | 0 | 0

9. Secondary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Marked Abnormality (Continued)
Description: ULN=upper limit of normal; LLN=lower limit of normal; BL=baseline. Creatine kinase (U/L), high:>5*ULN; protein, total(g/L):low if <0.90*BL when BL<LLN or <LLN when B >ULN or <0.90*LLN when BL is missing or LLN≤BL≤ULN, high if >1.10*BL if BL>ULN or >ULN when BL<LLN or >1.10*ULN if BL missing or LLN≤BL≤ULN.Protein,total(g/L): low if <0.90*BL if BL<LLN or <LLN if BL>ULN or <0.90*LLN if BL missing or LLN≤BL≤ULN, high if >1.10*BL if BL>ULN or >ULN if BL<LLN or >1.10*ULN if BL or LLN≤BL≤ULN; glucose, serum fasting (mg/dL): low if <0.8*BL if BL<LLN or <LLN when BL>ULN or <0.8*LLN when BL missing or LLN≤BL≤ULN, high if >2*BL when BL>ULN or >ULN when BL<LLN or >1.5*ULN if BL missing or LLN≤BL≤ULN; uric acid (mg/dL), high: >2*BL and BL>ULN or>1.5*ULN when BL missing or BL≤ULN; glucose, urine, high; protein, urine, high; blood, urine, high; leukocyte esterase, urine, high; RBC count, urine (Hpf), high; WBC count, urine (Hpf), high: ≥2 if BL=missing,=0 or =0.5 or if ≥3 if BL=1, or if ≥4 and BL≥2.
Time Frame: First dose of study drug (Day 1) to 30 days after last dose of blinded study drug
Population: Participants who received at least 1 dose of study drug. n=number evaluable
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily
Number analyzed (Participants) | 2798 | 2780
Participants
  Creatine kinase, low (n=2780, 2758) | 0 | 0
  Creatine kinase, high (n=2780, 2758) | 13 | 25
  Protein (total), low (n=103, 109) | 0 | 0
  Protein (total), high (n=103, 109) | 0 | 0
  Uric acid, low (n=386, 390) | 0 | 0
  Uric acid, high (n=386, 390) | 1 | 0
  Glucose (urine), low (n=2, 3) | 0 | 0
  Glucose (urine), high (n=2, 3) | 0 | 1
  Protein (urine), low (n=3, 5) | 0 | 0
  Protein (urine), high (n=3, 5) | 1 | 1
  Blood (urine), low (n=3, 5) | 0 | 0
  Blood (urine), high (n=3, 5) | 1 | 0
  Leukocyte esterase (urine), low (n=3,5) | 0 | 0
  Leukocyte esterase (urine), high (n=3,5) | 0 | 0
  Red blood cells (RBC) (urine), low (n=2,2) | 0 | 0
  RBC (urine), high (n=2,2) | 1 | 0
  White blood cells (urine), low (n=2,2) | 0 | 0
  WBC (urine), high (n=2,2) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 30 days (assessed up to May 2017, approximately 95 months)
Arm/Group | Apixaban, 2.5 or 5 mg Twice Daily | Acetylsalicylic Acid, 81-324 mg Once Daily | Open Label Apixaban
All-Cause Mortality (participants affected / at risk) | 111/2798 | 140/2780 | 286/3275
Serious Adverse Events (participants affected / at risk) | 657/2798 | 804/2780 | 1228/3275
Other Adverse Events (participants affected / at risk) | 207/2798 | 267/2780 | 180/3275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban, 2.5 or 5 mg Twice Daily (N=2798) | Acetylsalicylic Acid, 81-324 mg Once Daily (N=2780) | Open Label Apixaban (N=3275)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 11 | 19 | 25
Alcohol abuse (Psychiatric disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 7 | 6 | 8
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 1 | 10
Bronchitis (Infections and infestations) | 7 | 7 | 15
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 60 | 76 | 116
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 5
Cataract operation (Surgical and medical procedures) | 0 | 1 | 2
Cerebral infarction (Nervous system disorders) | 1 | 6 | 10
Chest pain (General disorders) | 16 | 24 | 28
Cholecystitis (Hepatobiliary disorders) | 5 | 6 | 4
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 1
Dengue fever (Infections and infestations) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 10 | 6
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 16
Eye haemorrhage (Eye disorders) | 2 | 0 | 0
Fasciotomy (Surgical and medical procedures) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 2 | 1
Gallbladder operation (Surgical and medical procedures) | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Genitourinary operation (Surgical and medical procedures) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 1 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 6 | 3 | 3
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 3 | 12
Infection (Infections and infestations) | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 2 | 1
Intermittent claudication (Vascular disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 2 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 1 | 6
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5 | 15
Malaise (General disorders) | 1 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 2 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 4 | 2 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 6
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Papilloma excision (Surgical and medical procedures) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 2
Peripheral nerve palsy (Nervous system disorders) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 2 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 3
Renal failure acute (Renal and urinary disorders) | 8 | 9 | 0
Septic shock (Infections and infestations) | 4 | 2 | 12
Skin graft (Surgical and medical procedures) | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 4
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 2 | 0 | 0
Wound infection (Infections and infestations) | 2 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 2
Abdominoplasty (Surgical and medical procedures) | 0 | 1 | 0
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 2 | 0
Atrioventricular block (Cardiac disorders) | 1 | 2 | 3
Bile duct stone (Hepatobiliary disorders) | 1 | 3 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 5 | 4 | 11
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 2 | 5 | 0
Cardiac pacemaker removal (Surgical and medical procedures) | 1 | 0 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 | 1 | 2
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 6 | 2
Device pacing issue (General disorders) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2 | 3
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 3
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 5 | 6 | 3
Gastritis erosive (Gastrointestinal disorders) | 1 | 2 | 2
Gout (Metabolism and nutrition disorders) | 2 | 2 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Hepatic amoebiasis (Infections and infestations) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 5
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 4
Implant site effusion (General disorders) | 0 | 1 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 6
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 3
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2 | 7
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Omentum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 4 | 4
Peptic ulcer (Gastrointestinal disorders) | 1 | 2 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic operation (Surgical and medical procedures) | 1 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Renal failure (Renal and urinary disorders) | 1 | 6 | 6
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2 | 0
Tarsal tunnel decompression (Surgical and medical procedures) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 1
Tracheitis (Infections and infestations) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 3 | 2 | 2
Ventricular failure (Cardiac disorders) | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 1 | 0
Abscess (Infections and infestations) | 0 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 2
Activities of daily living impaired (Social circumstances) | 0 | 1 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 12 | 11 | 23
Atrial fibrillation (Cardiac disorders) | 72 | 70 | 113
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 7
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 3 | 1 | 10
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 24
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 1 | 1
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 1
Device lead damage (General disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 22
Embolic stroke (Nervous system disorders) | 0 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 4 | 6 | 12
Femoral artery embolism (Vascular disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Generalised oedema (General disorders) | 1 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 2 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6
Haemorrhage (Vascular disorders) | 1 | 3 | 6
Hemiparesis (Nervous system disorders) | 1 | 1 | 0
Hernia pain (General disorders) | 0 | 1 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0
Implantable defibrillator replacement (Surgical and medical procedures) | 1 | 0 | 2
Inguinal hernia repair (Surgical and medical procedures) | 4 | 0 | 4
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 2
Lymphocele (Vascular disorders) | 1 | 0 | 0
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0 | 0
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 3 | 2 | 4
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1 | 0
Peripheral artery angioplasty (Surgical and medical procedures) | 1 | 1 | 3
Peripheral embolism (Vascular disorders) | 0 | 1 | 2
Physical assault (Social circumstances) | 1 | 0 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 5 | 2 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 1 | 8
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 2
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 5
Retinal detachment (Eye disorders) | 0 | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 1
Sinoatrial block (Cardiac disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Starvation (Metabolism and nutrition disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 2 | 0 | 0
Sudden cardiac death (General disorders) | 3 | 1 | 6
Supraventricular tachycardia (Cardiac disorders) | 3 | 5 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 1 | 0
Therapeutic embolisation (Surgical and medical procedures) | 1 | 0 | 0
Transfusion (Surgical and medical procedures) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 2
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Venous insufficiency (Vascular disorders) | 1 | 0 | 0
Vertebroplasty (Surgical and medical procedures) | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 6 | 7
Aortic rupture (Vascular disorders) | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 2 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 1 | 0
Arthritis bacterial (Infections and infestations) | 2 | 0 | 0
Asthenia (General disorders) | 4 | 1 | 9
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 2
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder mass (Renal and urinary disorders) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 2 | 0
Cardiac ablation (Surgical and medical procedures) | 1 | 2 | 1
Cardiac death (General disorders) | 1 | 1 | 3
Cardiac pacemaker insertion (Surgical and medical procedures) | 4 | 2 | 9
Cardiopulmonary failure (Cardiac disorders) | 2 | 3 | 4
Carditis (Cardiac disorders) | 0 | 1 | 0
Cerebral microhaemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral thrombosis (Nervous system disorders) | 1 | 0 | 0
Cervical root pain (Nervous system disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 4 | 6 | 16
Coronary artery insufficiency (Cardiac disorders) | 1 | 0 | 0
Cystoscopy (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 5 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 1 | 3
Epilepsy (Nervous system disorders) | 2 | 1 | 3
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 3 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 8 | 5 | 14
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 9 | 20
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 3 | 1 | 1
Haematuria (Renal and urinary disorders) | 5 | 4 | 13
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Hepatic enzyme increased (Investigations) | 1 | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 4 | 9 | 13
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 3 | 3 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 5
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Medical device complication (General disorders) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Orchidectomy (Surgical and medical procedures) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 6 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 3 | 17
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 3
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 2 | 2 | 0
Pneumonia (Infections and infestations) | 37 | 55 | 99
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 2 | 1 | 2
Pyelonephritis (Infections and infestations) | 1 | 0 | 2
Pyometra (Infections and infestations) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 8 | 11 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Thrombosis (Vascular disorders) | 1 | 1 | 1
Toe amputation (Surgical and medical procedures) | 0 | 1 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 4 | 1
Urethral disorder (Renal and urinary disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 3 | 3 | 4
Vertigo (Ear and labyrinth disorders) | 1 | 3 | 5
Angina unstable (Cardiac disorders) | 20 | 12 | 17
Angiogram (Investigations) | 1 | 3 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 3 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 39 | 28 | 53
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 3 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 1 | 1
Cellulitis (Infections and infestations) | 6 | 5 | 13
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 2 | 0
Coronary angioplasty (Surgical and medical procedures) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 3 | 0
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 5 | 6 | 11
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 2 | 1 | 8
Hip surgery (Surgical and medical procedures) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3 | 6
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 3
Ischaemic stroke (Nervous system disorders) | 19 | 46 | 22
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Lymph node cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 5 | 1 | 5
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 2 | 1 | 7
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Spigelian hernia (Gastrointestinal disorders) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 7
Systemic inflammatory response syndrome (General disorders) | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 10 | 29 | 13
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1 | 0 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 4
Ventricular fibrillation (Cardiac disorders) | 1 | 2 | 3
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 3
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 0 | 0
Angioplasty (Surgical and medical procedures) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 2 | 4
Arterial stenosis (Vascular disorders) | 0 | 1 | 0
Arteriogram coronary (Investigations) | 1 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 3 | 8
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 3 | 2 | 7
Clostridium colitis (Infections and infestations) | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Device malfunction (General disorders) | 0 | 1 | 0
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 3 | 7
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 2
Eye operation (Surgical and medical procedures) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 2
Gangrene (Infections and infestations) | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 4
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 5 | 6 | 8
Heart valve operation (Surgical and medical procedures) | 0 | 2 | 0
Hospitalisation (Surgical and medical procedures) | 3 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 2
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mastectomy (Surgical and medical procedures) | 0 | 1 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pelvic mass (General disorders) | 0 | 1 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Pneumonia viral (Infections and infestations) | 0 | 2 | 0
Renal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 5 | 6
Retinal artery embolism (Eye disorders) | 1 | 0 | 0
Salivary gland operation (Surgical and medical procedures) | 0 | 1 | 0
Sepsis (Infections and infestations) | 4 | 4 | 17
Shock (Vascular disorders) | 1 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 4
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 1
Thyroid haemorrhage (Endocrine disorders) | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 11 | 15 | 24
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 6
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Angina pectoris (Cardiac disorders) | 4 | 9 | 14
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 3
Aortic aneurysm (Vascular disorders) | 0 | 1 | 2
Aortic stenosis (Vascular disorders) | 2 | 0 | 3
Aphasia (Nervous system disorders) | 0 | 1 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 9
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5 | 12
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 2 | 1 | 3
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0
Bronchiectasis (Infections and infestations) | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 3 | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 7 | 10
Cardiac failure chronic (Cardiac disorders) | 0 | 3 | 6
Carotid arterial embolus (Nervous system disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 6
Cerebral cyst (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 5
Cor pulmonale (Cardiac disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 2 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 11
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 8
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 2 | 4
Heart rate irregular (Investigations) | 1 | 0 | 1
Hernia (General disorders) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 6 | 12
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 3 | 5
Mitral valve repair (Surgical and medical procedures) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 11 | 12 | 24
Oedema (General disorders) | 1 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 3 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 4 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 2 | 1
Pyrexia (General disorders) | 3 | 3 | 7
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Renal stone removal (Surgical and medical procedures) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Syncope (Nervous system disorders) | 8 | 18 | 26
Thromboembolectomy (Surgical and medical procedures) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 3
Urosepsis (Infections and infestations) | 1 | 1 | 4
Varicose vein (Vascular disorders) | 0 | 1 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Brain stem haemorrhage (Nervous system disorders) | 0 | 1 | 0
Bursal operation (Surgical and medical procedures) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 3 | 7 | 3
Cardioversion (Surgical and medical procedures) | 1 | 0 | 0
Cerebellar ataxia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 16 | 40 | 15
Cholangitis (Hepatobiliary disorders) | 2 | 0 | 3
Cholecystitis acute (Hepatobiliary disorders) | 5 | 2 | 4
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Death (General disorders) | 14 | 9 | 38
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 4 | 6
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Hernia repair (Surgical and medical procedures) | 1 | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 5 | 4 | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 4 | 4
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Incisional hernia repair (Surgical and medical procedures) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 3 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 1
Liver function test abnormal (Investigations) | 1 | 2 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Microvascular angina (Cardiac disorders) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 3 | 5 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 3 | 5 | 3
Peripheral ischaemia (Vascular disorders) | 0 | 5 | 3
Phlebitis (Vascular disorders) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 10 | 12
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal polypectomy (Surgical and medical procedures) | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Splenic artery aneurysm (Gastrointestinal disorders) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 2 | 5
Sudden death (General disorders) | 9 | 12 | 32
Swelling (General disorders) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Dementia alzheimer's type (Nervous system disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1
Hyponatraemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 0 | 1
Neuritis (Nervous system disorders) | 0 | 0 | 1
Neuroglycopenia (Nervous system disorders) | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 3
Simple partial seizures (Nervous system disorders) | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 1
Subdural effusion (Nervous system disorders) | 0 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 1
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 0 | 1
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Lead dislodgement (Product Issues) | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1
Bipolar i disorder (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 24
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 2
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 3
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2
Postrenal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatic hypoplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 2
Spermatic cord disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Cardiac assistance device user (Social circumstances) | 0 | 0 | 1
Aortic aneurysm repair (Surgical and medical procedures) | 0 | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 0 | 1
Benign tumour excision (Surgical and medical procedures) | 0 | 0 | 1
Bladder polypectomy (Surgical and medical procedures) | 0 | 0 | 1
Cancer surgery (Surgical and medical procedures) | 0 | 0 | 1
Carotid endarterectomy (Surgical and medical procedures) | 0 | 0 | 2
Choledochoenterostomy (Surgical and medical procedures) | 0 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 0 | 2
Endarterectomy (Surgical and medical procedures) | 0 | 0 | 1
Endovenous ablation (Surgical and medical procedures) | 0 | 0 | 1
Gastric bypass (Surgical and medical procedures) | 0 | 0 | 1
Gastrointestinal tube insertion (Surgical and medical procedures) | 0 | 0 | 1
Heart valve replacement (Surgical and medical procedures) | 0 | 0 | 1
High frequency ablation (Surgical and medical procedures) | 0 | 0 | 1
Hydronephrosis repair (Surgical and medical procedures) | 0 | 0 | 1
Knee operation (Surgical and medical procedures) | 0 | 0 | 1
Laparotomy (Surgical and medical procedures) | 0 | 0 | 1
Liver operation (Surgical and medical procedures) | 0 | 0 | 1
Lung operation (Surgical and medical procedures) | 0 | 0 | 1
Medical device implantation (Surgical and medical procedures) | 0 | 0 | 1
Medical device removal (Surgical and medical procedures) | 0 | 0 | 1
Mitral valve replacement (Surgical and medical procedures) | 0 | 0 | 1
Pancreaticoduodenectomy (Surgical and medical procedures) | 0 | 0 | 1
Plastic surgery to the face (Surgical and medical procedures) | 0 | 0 | 1
Proctocolectomy (Surgical and medical procedures) | 0 | 0 | 1
Rehabilitation therapy (Surgical and medical procedures) | 0 | 0 | 1
Skin lesion removal (Surgical and medical procedures) | 0 | 0 | 1
Thyroid operation (Surgical and medical procedures) | 0 | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 0 | 1
Tracheostomy (Surgical and medical procedures) | 0 | 0 | 1
Ureteral stent insertion (Surgical and medical procedures) | 0 | 0 | 1
Urethral stent insertion (Surgical and medical procedures) | 0 | 0 | 1
Vascular graft (Surgical and medical procedures) | 0 | 0 | 1
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 0 | 0 | 1
Weight loss diet (Surgical and medical procedures) | 0 | 0 | 1
Wrist surgery (Surgical and medical procedures) | 0 | 0 | 1
Unassigned (General disorders) | 4 | 6 | 7
Accelerated hypertension (Vascular disorders) | 0 | 0 | 1
Aneurysm (Vascular disorders) | 0 | 0 | 1
Arterial disorder (Vascular disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 2
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 2
Leriche syndrome (Vascular disorders) | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 0 | 1
Varicose ulceration (Vascular disorders) | 0 | 0 | 1
Varicose vein ruptured (Vascular disorders) | 0 | 0 | 1
Venous haemorrhage (Vascular disorders) | 0 | 0 | 1
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Cardiac asthma (Cardiac disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 3
Defect conduction intraventricular (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 2
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 4
Nodal rhythm (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1
Rheumatic heart disease (Cardiac disorders) | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 0 | 2
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 18
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Liddle's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 2
Eyelid ptosis (Eye disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1
Tolosa-hunt syndrome (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 3
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 3
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal dilatation (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 14
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 0 | 1
Incarcerated hernia (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 5
Peripheral swelling (General disorders) | 0 | 0 | 1
Unevaluable event (General disorders) | 0 | 0 | 2
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 2
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis fulminant (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Abdominal wall infection (Infections and infestations) | 0 | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 2
Diabetic foot infection (Infections and infestations) | 0 | 0 | 2
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 0 | 2
Empyema (Infections and infestations) | 0 | 0 | 1
Encephalitis viral (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 8
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 3
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Groin infection (Infections and infestations) | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Listeriosis (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Prostate infection (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 2
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aortic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 2
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stomal hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 5
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arthroscopy (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 1
Ecg signs of myocardial ischaemia (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 2
Heart rate abnormal (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
B-cell small lymphocytic lymphoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Light chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 4
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 2
Cerebral artery embolism (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban, 2.5 or 5 mg Twice Daily (N=2798) | Acetylsalicylic Acid, 81-324 mg Once Daily (N=2780) | Open Label Apixaban (N=3275)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 109 | 141 | 164
Dizziness (Nervous system disorders) | 109 | 144 | 132

LIMITATIONS AND CAVEATS:
On May 28, 2010, after a planned interim analysis for efficacy, the Data Monitoring Committee recommended early termination due to apixaban's superior efficacy over ASA, with an acceptable safety profile. The open-label phase is ongoing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.